CLINICAL TRIAL: NCT00917449
Title: Interventional Pharmacological Study With L-Arginine in the Prevention of Type 2 Diabetes Mellitus in Patients With Metabolic Syndrome
Brief Title: Prevention of Type 2 Diabetes Mellitus by L-Arginine in Patients With Metabolic Syndrome
Acronym: L-arginine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Piatti PierMarco, San Raffaele Scientific Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2005-004639-24
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Metabolic Syndrome; Impaired Glucose Tolerance; Insulin Resistance; Endothelial Dysfunction
Keywords: Metabolic Syndrome; Impaired glucose tolerance; Type 2 diabetes mellitus; Endothelial dysfunction; L-arginine; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-arginine (Active Comparator): L-arginine (3.2 gr bid) plus lifestyle counselling vs placebo plus lifestyle counselling
  Interventions: Drug: L-arginine
- placebo (Placebo Comparator): placebo plus lifestyle counselling for 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-arginine — Oral L-arginine (3.2 gr bid)for 18 months
  Other Names: bioarginine
  Arms: L-arginine
Drug: Placebo — Oral Placebo BID for 18 months
  Arms: placebo

SUMMARY:
Aim

The principal objective of this project is:

• To evaluate the efficacy of long term (18 months) L-Arginine therapy in preventing or delaying clinical onset of type 2 diabetes mellitus in subjects with impaired glucose tolerance (IGT) and Metabolic Syndrome.

Secondary end points are:

1. To define if a long term treatment with L-arginine is able to ameliorate insulin sensitivity and endothelial dysfunction in this population.
2. To find new risk profiles and candidate genes able to define the sub-group of patients at higher risk to develop type 2 diabetes mellitus.

Methodology This is a double blind, parallel, one centre study to determine if long term oral L-arginine administration is able to delay or prevent type 2 diabetes mellitus in patients with Metabolic Syndrome. Two hundred and ninety four subjects were recruited at the Cardio-Metabolic and Clinical Trials Unit of the San Raffaele Scientific Institute. One hundred and forty two patients were randomized to enter the study and assigned to two arms: oral L-arginine (6.4 g/die) or placebo, in addition to diet and physical exercise. The treatment were maintained for 18 months. Visits were performed every 3 months for clinical evaluation, blood samples, treatment supply and collection of data on adverse events. Furthermore, patients were contacted every month by telephone to evaluate the accurate continuation of the study and they were instructed to phone to the centre in case of possible adverse events.

An OGTT were performed before the enter into the study and at the end of the study period. An additional OGTT were performed at an intermediate visit if fasting glucose levels were more than 126 mg/dl. A diabetic response caused the end-point of the patient. Metabolic, hormonal and endothelial activation and inflammation parameters were measured. Evaluation of endothelium-mediated and non-endothelium-mediated vasodilatation were performed by strain gauche plethysmography evaluating forearm blood at the basal state. in post-ischemic conditions and after nitroglycerine administration.

Before the enter into the study, an additional blood sample were drawn for DNA extraction and candidate genes variants evaluation. Before the enter into the study and at the end of the study period, gene expression for inflammation were measured on mRNA extraction on endothelial progenitor cells.

DETAILED DESCRIPTION:
This is a double blind, parallel, one centre study to determine if long term oral L-arginine administration is able to delay or prevent type 2 diabetes mellitus in patients with IGT and Metabolic Syndrome. Two hundred and ninety four subjects were recruited at the CardioMetabolic and Clinical Trials Unit of the San Raffaele Scientific Institute. One hundred and fourty two patients were randomized to enter the study. Patients were randomly assigned to two arms: oral L-arginine (6.4 g/die) or placebo in blind scheme. The treatment were maintained for 18 months. Visits will be performed every 3 months for clinical evaluation, blood samples, treatment supply and collect data on adverse events, if any. Furthermore, patients were contacted every month by telephone to evaluate the accurate continuation of the study and they were instructed to phone to the centre in case of possible adverse events.

Inclusion criteria

* Written informed consent must be obtained before any procedure of the study is done.
* Male or Female aged more than 35 years.
* Diagnosis of IGT after a standard Glucose Tolerance Test (OGTT, 75 g)
* Moreover, in order to be considered affected by Metabolic Syndrome, they must have two or more of the following criteria:
* Abdominal obesity (waist>120 cm for man, >88 cm for women)
* Hypertriglyceridemia (>150 mg/dl)
* Low HDL cholesterol (<40mg/dl in man, <50 mg/dl in woman)
* Hypertension (>130 / >85 mmHg) Exclusion criteria
* Presence of type 1 or type 2 diabetes mellitus
* Fasting glucose levels >126 mg/dl
* Sitting Systolic Arterial Pressure >140mmHg, and Sitting Diastolic Arterial Pressure >90mmHg
* Pregnancy
* Known renal insufficiency or creatinine levels more than 1.8 mg/dl,
* Presence of chronic hepatopathy or levels of ALT and AST more than two standard deviations from normality levels
* Presence of malignancy
* Abuse of alcohol or abuse substances
* Psychiatric disorders

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any procedure of the study is done.
* Male or Female aged more than 35 years.
* Diagnosis of IGT after a standard Glucose Tolerance Test (OGTT, 75 g)
* Moreover, in order to be considered affected by Metabolic Syndrome, they must have two or more of the following criteria:
* Abdominal obesity (waist>120 cm for man, >88 cm for women)
* Hypertriglyceridemia (>150 mg/dl)
* Low HDL cholesterol (<40mg/dl in man, <50 mg/dl in woman)
* Hypertension (>130 / >85 mmHg)

Exclusion Criteria:

* Presence of type 1 or type 2 diabetes mellitus
* Fasting glucose levels >126 mg/dl
* Sitting Systolic Arterial Pressure >140mmHg, and Sitting Diastolic Arterial Pressure >90mmHg
* Pregnancy
* Known renal insufficiency or creatinine levels more than 1.8 mg/dl,
* Presence of chronic hepatopathy or levels of ALT and AST more than two standard deviations from normality levels
* Presence of malignancy
* Abuse of alcohol or abuse substances
* Psychiatric disorders

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of long term (18 months) L-Arginine therapy in preventing or delaying clinical onset of type 2 diabetes mellitus in subjects with impaired glucose tolerance (IGT) and Metabolic Syndrome. | 18 months

SECONDARY OUTCOMES:
Define if the treatment with L-arginine can ameliorate insulin sensitivity and endothelial dysfunction and find new risk profiles and candidate genes able to characterize the sub-group of patients at higher risk to develop type 2 diabetes mellitus. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: PierMarco Piatti, MD, Principal Investigator — Scientific Institute San Raffaele
Locations (1):
- Scientific Institute San Raffaele, Milan, Milan, Italy

REFERENCES:
- [Derived] Monti LD, Galluccio E, Villa V, Fontana B, Spadoni S, Piatti PM. Decreased diabetes risk over 9 year after 18-month oral L-arginine treatment in middle-aged subjects with impaired glucose tolerance and metabolic syndrome (extension evaluation of L-arginine study). Eur J Nutr. 2018 Dec;57(8):2805-2817. doi: 10.1007/s00394-017-1548-2. Epub 2017 Oct 20. PMID 29052766
- [Derived] Monti LD, Galluccio E, Fontana B, Spadoni S, Comola M, Marrocco Trischitta MM, Chiesa R, Comi G, Bosi E, Piatti P. Pharmacogenetic influence of eNOS gene variant on endothelial and glucose metabolism responses to L-arginine supplementation: Post hoc analysis of the L-arginine trial. Metabolism. 2015 Nov;64(11):1582-91. doi: 10.1016/j.metabol.2015.08.015. Epub 2015 Aug 28. PMID 26385052